CLINICAL TRIAL: NCT02582554
Title: Efficacy of Nutrition Risk Screening With NutriSTEP® in Toddlers and Preschoolers
Acronym: NutriSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Janis Randall Simpson, College Professor Emerita, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 052454
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Dietary Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention: NutriSTEP The intervention will be the administration of NutriSTEP, a nutrition risk screening questionnaire for preschoolers along with a nutrition education brochure called How to Build a Healthy Preschooler
  Interventions: Behavioral: NutriSTEP
- Control (No Intervention): Control: Wait-list control The wait-list control group will complete the NutriSTEP and receive the nutrition education information at the end of the 3 month study period

INTERVENTIONS:
Behavioral: NutriSTEP — Provision of nutrition risk screening with NutriSTEP (a nutrition risk screening questionnaire for preschoolers) and nutrition education with NutriSTEP related materials
  Other Names: How to Build a Healthy Preschooler
  Arms: Intervention

SUMMARY:
Good nutrition is necessary for optimal growth and development in young children. Nutrition risk screening can identify those at risk and to refer them for assessment and treatment. The NutriSTEP® (Nutrition Risk Screening for Every Preschooler) questionnaires are 17-item, community-based, parent-administered questionnaires for identifying nutritional risk in toddlers (18-35 months) and preschoolers (3-5 years). Internet versions are available on the Dietitians of Canada website as part of a Nutri-eSTEP online tool. NutriSTEP® is mandated for use in Ontario and New Brunswick and is also used in other provinces. NutriSTEP® has been implemented in Canadian jurisdictions and in research settings. Many health care practitioners, mainly registered dietitians, and policy makers, are asking for evidence that NutriSTEP® makes a difference and this project is proposed to show that nutrition screening with NutriSTEP® with its accompanying nutrition education resources will increase knowledge and change nutrition-related practices by parents of preschoolers.

This research will be a randomized control trial with more than 150 parents/caregivers of toddlers and preschoolers. The treatment group will receive screening with the Nutri-eSTEP version of NutriSTEP® and will receive the accompanying nutrition education messages and links to resources. A control group will receive the screening treatment at the end of a 12 week intervention. At the beginning and end of the 12 week period, parents/caregivers will fill out questionnaires on parental nutrition knowledge and nutrition-related behaviour (including attitudes and intentions).

This will be the first study of nutrition risk screening with NutriSTEP® to determine if the screening process, along with its accompanying nutrition education messages makes a difference.

DETAILED DESCRIPTION:
Study Design The proposed research will be a wait-listed randomized control trial of the efficacy of the NutriSTEP® screening process for toddlers and preschoolers. The treatment group will undergo screening with Nutri-eSTEP plus its accompanying nutrition education messages and links to resources. A control group will be wait-listed to receive the treatment (Nutri-eSTEP plus its accompanying nutrition education treatment) at the end of the intervention period.

Outcome variables Participants Parents/caregivers of toddlers and preschoolers will be recruited at various Ontario Early Years Centres (OEYCs) in southern Ontario.

Sample Size The sample size (http://www.stat.ubc.ca/) is estimated at 63 per group based on difference in scores on the NKQ of 2 (~half of the difference found between students and parents), with a SD of 4, alpha of 0.05 and statistical power of 0.80 (2-tailed). An allowance for 20% attrition (based on our previous test-retest reliability studies)(7,8,19) will see 77 participants per group recruited. This will also allow for enough power for an improvement in NutriSTEP® scores based on a difference of 2.2 units, standard deviation of 5, alpha of 0.05 and statistical power of 0.80 (1-tailed)(based on a difference in NutriSTEP® scores over 3 months of a parenting intervention study (56). The total sample of 154 will be recruited from ~20 OEYCs @ ~10 participants/site (based on previous experience).

Intervention NutriSTEP® Questionnaire: The toddler and preschool NutriSTEP® questionnaires will form part of the intervention for this trial.

Nutrition Education Material:

"How to Build a Healthy Toddler/Preschooler": This booklet will be part of the intervention for this trial. "How to Build a Healthy Toddler/Preschooler" are 4-page brochures that have key messages relevant to the questions on the NutriSTEP® questionnaires. Recommendations from Canada's Food Guide (CFG) are included as well as suggestions for credible nutrition resources.

Nutri-eSTEP Feedback Messages: As part of the Nutri-eSTEP platform, parents receive feedback messages based on their responses to each question on the NutriSTEP®. The feedback messages are categorized into two categories: "What is Going Well" and "What to Work On". For this study, we will provide print copies of the Results and feedback messages to participants as part of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of 3-5 year old children, speak English, read English at Grade 6 level

Exclusion Criteria:

* Parent of an institutionalized child

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Score of Nutritional Risk as Assessed by the NutriSTEP Nutrition Knowledge Questionnaire | 12 weeks
  A valid and reliable 40-item nutrition knowledge questionnaire has been developed to test the contents of the NutriSTEP questionnaire and its accompanying nutrition education material. Correct scores on the items on the questionnaire will be added up for a total score, with differences between the start of the study and the end of the study compared and also a comparison between the intervention and control groups.

SECONDARY OUTCOMES:
Score of Nutrition Behaviour as Assessed by the NutriSTEP Questionnaire | 12 weeks
  The NutriSTEP Behaviour Questionnaire is a valid and reliable 17-item questionnaire to assess nutrition-related behaviours in preschoolers. Each response item for the 17 questions is assigned a score. Total scores will be generated, with comparisons at the start and end of the study and between the intervention and control groups.
Score of Attitudes and Self-Efficacy as Determined by the NutriSTEP Attitudes and Self-Efficacy Questionnaire | 12 weeks
  A valid and reliable 21-item questionnaire to assess attitudes and self-efficacy related to the NutriSTEP questionnaire has been developed. Response categories for each item on each of the attitudes and self-efficacy questions are scored. Scores are added up for each of the attitudes and self-efficacy portions of the questionnaire. Differences between scores before and after the intervention and between intervention and control groups will be compared.
Score of Intentions to Change Behaviour as Determined by the NutriSTEP Intentions Questionnaire | 12 weeks
  The NutriSTEP Intentions Questionnaire is a valid and reliable 7-item questionnaire. A total score is generated based on the scores for the response categories for each item on the questionnaire. Differences in scores between the start of the study and the end of the study and also between the intervention and the control groups will be determined.